CLINICAL TRIAL: NCT03487848
Title: Open-Label, Single-Arm Trial to Evaluate the Pharmacokinetics, Safety and Efficacy of Daclatasvir (DCV) in Combination With Sofosbuvir (SOF) in Children From 3 to Less Than 18 Years of Age With GT-1 to -6 Chronic Hepatitis C (CHC) Infection
Brief Title: Evaluation of Daclatasvir (DCV) in Combination With Sofosbuvir (SOF) in Children With Chronic Hepatitis C (CHC) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-423; 2017-003338-94 (EudraCT Number)
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C; Chronic Hepatitis
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic | interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Daclatasvir with Sofosbuvir (Experimental): Specified dose on specified days for specified duration
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir — Specified dose on specified days for specified duration
Drug: Sofosbuvir — Specified dose on specified days for specified duration

SUMMARY:
The purpose of this study is to evaluate daclatasvir in combination with sofosbuvir given to children with chronic hepatitis C infection

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants monoinfected with HCV genotype -1 to -6
* HCV RNA ≥1,000 IU/mL at Screening
* Participants who are HCV-treatment naïve or treatment experienced
* Participants in Cohort 1 must have a body weight ≥ 45kg at Day 1

Exclusion Criteria:

* Mixed genotype HCV infections
* Evidence of an ongoing medical condition contributing to chronic liver disease other than HCV
* Evidence of cirrhosis, either compensated or decompensated
* Prior exposure to sofosbuvir and/or NS5A inhibitor

Other protocol defined inclusion/exclusion criteria could apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Melbourne, Victoria, Australia
- Local Institution, Barcelona, Spain

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were enrolled and treated
Groups:
- Daclatasvir (DCV) + Sofosbuvir (SOF): DCV 60 mg QD + SOF 400 mg QD for 12 weeks
Period: Overall Study
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Minimum (Trough) Observed Plasma Concentration (Cmin) for Daclatasvir
Time Frame: Day 10 after first dose, collection timepoints at pre-dose, 30 min, 1 hour, 2 hours, 4 hours, and 8 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
ng/mL | 152.94 (48.3)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Daclatasvir
Time Frame: Day 10 after first dose, collection timepoints at pre-dose, 30 min, 1 hour, 2 hours, 4 hours, and 8 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
ng/mL | 1215.32 (37.2)

3. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) for Daclatasvir
Time Frame: Day 10 after first dose, collection timepoints at pre-dose, 30 min, 1 hour, 2 hours, 4 hours, and 8 hours post-dose
Population: All treated participants
Measure: Median (Full Range); unit: Hours
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Hours | 2.00 [1.0 to 4.0]

4. Primary Outcome: Area Under the Concentration-Time Curve (AUC(TAU)) for Daclatasvir
Time Frame: Day 10 after first dose, collection timepoints at pre-dose, 30 min, 1 hour, 2 hours, 4 hours, and 8 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
h*ng/mL | 11535.45 (26.6)

5. Primary Outcome: Apparent Total Body Clearance (CLT/F) for Daclatasvir
Time Frame: Day 10 after first dose, collection timepoints at pre-dose, 30 min, 1 hour, 2 hours, 4 hours, and 8 hours post-dose
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
mL/min | 86.69 (22.3)

6. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: This outcome describes the number of participants experiencing different types of any grade adverse events.
Time Frame: From first dose to last dose (12 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Participants
  Adverse Events (AEs) | 4
  Serious Adverse Events (SAEs) | 0
  AEs leading to discontinuation | 0

7. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities - On-treatment Analysis
Description: Laboratory tests abnormalities were analyzed in the following categories:
  * Hematology (hemoglobin, platelets, international normalized ratio (INR), white blood cell count (WBC), lymphocytes (absolute), neutrophils + bands (absolute; ANC)).
  * Hepatobiliary enzymes (ALT, AST, alkaline phosphatase, total bilirubin, albumin).
  * Pancreatic enzymes (lipase, creatinine). Tests results were reported by worst toxicity grade (0 to 4) based on the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (2017).
  Only laboratory abnormalities with a worst toxicity grade 3 or higher in any of the above-mentioned tests, experienced during the on-treatment period, are reported here.
Time Frame: From the day after first dose to last dose (approximately 12 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Participants | 1

8. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities - Follow-up Analysis
Description: Laboratory tests abnormalities were analyzed in the following categories:
  * Hematology (hemoglobin, platelets, international normalized ratio (INR), white blood cell count (WBC), lymphocytes (absolute), neutrophils + bands (absolute; ANC)).
  * Hepatobiliary enzymes (ALT, AST, alkaline phosphatase, total bilirubin, albumin).
  * Pancreatic enzymes (lipase, creatinine). Tests results were reported by worst toxicity grade (0 to 4) based on the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (2017).
  Only laboratory abnormalities with a worst toxicity grade 3 or higher in any of the above-mentioned tests, experienced during the follow-up period, are reported here.
Time Frame: From day after last dose to end of follow-up period (up to approximately 96 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Participants | 2

9. Secondary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) RNA Levels Below the Lower Limit of Quantitation (LLOQ) at Post-Treatment Follow-Up Week 12
Description: HCV RNA levels were measured by using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test v2.0. This assay has a lower limit of quantitation (LLOQ) = 15 IU/mL.
  The outcome includes both results where Target was Detected (TD) but below LLOQ and results were Target was Not Detected (TND)
Time Frame: 12 weeks after last dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
Number analyzed (Participants) | 5
Percent of Participants | 100 [50 to 100]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days following last dose
Arm/Group | Daclatasvir (DCV) + Sofosbuvir (SOF)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir (DCV) + Sofosbuvir (SOF) (N=5)
Abdominal pain (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early by sponsor for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03487848/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT03487848/SAP_001.pdf